CLINICAL TRIAL: NCT04138745
Title: Transverse Thoracic Plane Block in the Pediatric Cardiac Patient
Acronym: TTPPCT
Status: Completed | Type: Observational
Sponsor: Ochsner Health System (Other)
Responsible Party: Principal Investigator, Dominic Carollo, Senior Staff Physician, Ochsner Health System
Other Study IDs: TTP Peds Cardiac
Record Dates: First submitted 2019-10-23; First posted 2019-10-24 (Actual); Last update posted 2021-09-09 (Actual); Status verified 2021-09

CONDITIONS: Pain, Acute; Congenital Heart Disease
MeSH Terms: conditions — Acute Pain; Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control: Historical control patients that are matched to the surgery type
- Experimental: After the practice change of TTP was initiated, the future pediatric patients were put into a database.
  Interventions: Other: Transverse Thoracic Plane Block

INTERVENTIONS:
Other: Transverse Thoracic Plane Block — A bilateral plane block in the transverse thoracic space
  Groups: Experimental

SUMMARY:
Postoperative pain after cardiothoracic surgery can be a significant problem interfering with recovery, yet difficult to manage due to the sedating effects of opiates. These patients frequently have associated postoperative pulmonary changes and are at risk of respiratory depression with opioid analgesia. The ultrasound-guided transversus thoracic muscle plane block (TTMPB) is a recently described regional anesthetic technique showing improvements in postoperative pain management. Further investigation is needed to establish the potential of the TTMPB as an analgesic modality in congenital cardiothoracic surgery in patients under the age of 18.

ELIGIBILITY:
Inclusion Criteria:

* Congenital Heart Surgery

Exclusion Criteria:

* Over 18

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: All comers int he age groups above
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Extubation | 2 years
  The amount of time until the patients are extubated in the ICU or OR.

SECONDARY OUTCOMES:
Surgical Stress Response | 2 years
  HR response to incision
Opiate Usage | 2 years
  Amount of total opiates used for the heart surgery

CONTACTS AND LOCATIONS:
Overall Officials: DOMINIC S CAROLLO, MD, Principal Investigator — Ochsner Health System
Locations (1):
- Ochsner Health System, New Orleans, Louisiana, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP